CLINICAL TRIAL: NCT02847858
Title: Health-E You: Reducing Unintended Pregnancies Among Hispanic Adolescents Using a Computer-based Intervention
Brief Title: Health-E You: Reducing Unintended Pregnancies Among Hispanic Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kathleen Tebb, Prinicipal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AD-1502-27481
Record Dates: First submitted 2016-06-29; First posted 2016-07-28 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Unprotected Sex; Unsafe Sex
Keywords: unsafe sex; unprotected sex; adolescents; Latinas; Hispanic; mobile health applications; unintended pregnancy; teen pregnancy prevention; school-based health centers
MeSH Terms: conditions — Unsafe Sex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health-E You App Participants (Experimental)
  Interventions: Behavioral: Health-E You: a computer-based intervention to improve the use of effective contraception among Hispanic adolescents
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Health-E You: a computer-based intervention to improve the use of effective contraception among Hispanic adolescents — School-based health centers which were randomized into the intervention arm will use the Health-E You App (n=7 clinics).
  Arms: Health-E You App Participants

SUMMARY:
Health -E-You is an interactive, individually tailored computer application (App) that was developed to educate adolescent girls about contraceptive methods and assist them in selecting a contraceptive method that meets their individual needs. The goal is to reduce disparities in unintended pregnancy rates among Hispanic adolescent females.

The App was designed in close collaboration with clinicians and Hispanic adolescents. Health-E You was designed to be used in conjunction with a clinical encounter to prime both the patient and provider prior to the face-to-face visit to facilitate the discussion and provision of appropriate contraception. It is founded on key principles of Social Cognitive Theory.

Through an interactive approach, Health-E-You assesses the users' sexual health risks, knowledge and contraceptive use history and preferences to facilitate a sense of agency and self-efficacy around selecting an effective contraceptive method. First, the user selects their preferred language (English or Spanish) and according to the selected language, the App provides a brief description of the module and consents the user to participate. It then assesses sexual health knowledge using an interactive truth vs. myth game. Correct answers to the truth vs. myth statements are then presented to the user as short, easy-to-read explanations. Next, the App assesses the user's individual contraceptive needs and preferences. The user is also screened for possible medical contraindications to contraceptive methods. Based on the user's input, the App provides individually tailored messaging and recommendations for contraceptive methods according to the user's own timeline for childbearing and their lifestyle preferences, past experiences and needs. The recommendations are presented on a visual continuum of effective contraceptive options based on desired duration of action and efficacy. Users then have the option to learn more about the recommended method(s) and they also have the option to learn more about any of the contraceptive options. Evidence-based contraceptive information is presented in a user-friendly format that includes YouTube style videos. Users can select to view brief video vignettes that feature clinicians who provide additional information about the method of interest and/or videos of diverse young women who discuss their experiences with each of the contraceptive methods. At the end of the App, adolescents are asked to select the method (s) they are most interested in using. They are also encouraged to use condoms to protect against sexually transmitted infections (STIs) and provided information about emergency contraception. Users can review a summary of a key information gathered from the App and are offered the opportunity to share that information with their clinician so that the clinician can better support the adolescent in selecting and using an effective and appropriate contraceptive method.

The objective of this study is to evaluate the effectiveness of Health-E You on its ability to address disparities in contraceptive knowledge, access and utilization among Hispanic adolescents. The long term goal is to reduce the incidence of unprotected sexual intercourse (and associated unintended pregnancies and STIs) over time. A total of 14 School-Based Health Centers (SBHCs) affiliated with the Los Angeles Unified School District, will be randomized, with equal chance, to use the Health-E You App or to provide usual care (without the App). A total of 1400 Hispanic adolescents will be selected to participate in the study (700 at intervention clinics and 700 at the control clinics). The investigators hypothesize that adolescents who use the Health-E You App will have greater sexual health knowledge and will be more likely to use effective contraceptive than adolescent who do not use the App. The investigators will also evaluate the effectiveness of the App on its ability to improve the effectiveness and efficiency of the health visit. Participants will be asked to complete follow-up surveys immediately following the clinical encounter and at three and six months after the clinical encounter.

The ultimate goal of this study is address health disparities in the use of effective contraceptives and ultimately reduce the incidence of unintended pregnancies and STIs among at-risk Hispanic adolescent girls.

ELIGIBILITY:
Inclusion Criteria:

Female 14-18 years of age Hispanic/Latina English or Spanish-speaker Has had sexual intercourse

Exclusion Criteria:

Currently pregnant Currently using an intrauterine device or implant contraceptive method Male Under 14 or over 19 years of age Not sexually active Non-Hispanic / Latina

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1360 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Tebb, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Belmont Wellness Center, Los Angeles, California
  - Carson Wellness Center, Los Angeles, California

REFERENCES:
- [Derived] Tebb KP, Leng Trieu S, Rico R, Renteria R, Rodriguez F, Puffer M. A Mobile Health Contraception Decision Support Intervention for Latina Adolescents: Implementation Evaluation for Use in School-Based Health Centers. JMIR Mhealth Uhealth. 2019 Mar 14;7(3):e11163. doi: 10.2196/11163. PMID 30869649
- [Derived] Tebb KP, Rodriguez F, Pollack LM, Trieu SL, Hwang L, Puffer M, Adams S, Ozer EM, Brindis CD. Assessing the effectiveness of a patient-centred computer-based clinic intervention, Health-E You/Salud iTu, to reduce health disparities in unintended pregnancies among Hispanic adolescents: study protocol for a cluster randomised control trial. BMJ Open. 2018 Jan 10;8(1):e018201. doi: 10.1136/bmjopen-2017-018201. PMID 29326184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited from 18 participating school-based health centers in the Los Angeles UnifiedSchool District starting August 2016 and ending May 31, 2018. Clinic staff provided all female youth who entered the clinic an opportunity to use the iPad with the intervention app (baseline questionnaire for the control group).
Groups:
- Health-E You Intervention Arm: Intervention arm. Participants answered baseline questions and received individually-tailored contraception and reproductive health information from a web-based computer application on an iPad at one of the 9 school-based health centers that was randomized to the intervention arm.
- Control Arm: Control Arm. Participants in this arm of the study completed an online baseline questionnaire about their demographic information and sexual and reproductive health behavior on an iPad at one of the 9 school-based health centers randomly assigned to the control arm.
Period: Overall Study
Arm/Group | Health-E You Intervention Arm | Control Arm
Started | 693 | 667
Completed | 292 | 398
Not Completed | 401 | 269
Not completed — Lost to Follow-up | 401 | 269

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health-E You Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 693 | 667 | 1360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 693 | 667 | 1360
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — All data was collected using a mobile tablet in a study site. All information was self-reported by participants.
  Participants
    Female | 693 | 667 | 1360
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 693 | 667 | 1360
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 4 | 10
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 6 | 6 | 12
  Black or African American | 24 | 20 | 44
  White | 24 | 17 | 41
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 623 | 614 | 1237
Region of Enrollment [Number; unit: participants]
  United States | 693 | 667 | 1360
Reason for visit related to reproductive health services [Count of Participants; unit: Participants] — Did the participant visit the clinic for reproductive health or birth control related services.
  Data was collected on a mobile tablet device in the clinic as a part of a survey.
  Participants
    Visit related to reproductive health services | 550 | 349 | 899
    Visit not related to reproductive health services | 137 | 306 | 443
    Missing data | 6 | 12 | 18
Had sex in the past 3 months [Count of Participants; unit: Participants] — Participants indicated whether or not they had sex in the past 3 months in the Baseline, 3-Month, and 6-Month online surveys.
  Participants
    Yes had sex in past 3 months at Baseline | 586 | 504 | 1090
    No did not have sex in past 3 months at Baseline | 107 | 147 | 254
    Missing data | 0 | 16 | 16

OUTCOME MEASURES:

1. Primary Outcome: Contraception Use Self-efficacy Scale Score (Aim 1b)
Description: The 3-item attitude scale assessing perceived ability to choose and use contraception was self-administered in an online survey; each item scored on a 0=not at all confident to 10=completely confident scale; scale score is the sum of the 3 items scores, range 0 - 30 (higher score=greater self-efficacy)
Time Frame: Pre-visit Baseline, Post-visit Follow-up (48 hours after Baseline)
Population: All participants for whom a self-efficacy score was recorded either at Baseline or at Post-visit Follow-up
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Intervention: Used Health-E You app in waiting room prior to clinical visit
- Control: Usual care (app not offered)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 690 | 640
Scores on a scale
  Pre-visit Baseline | 23.2 (6.34) | 22.45 (6.72)
  Post-visit Follow-up (48 hours post Baseline): number analyzed (Participants) | 320 | 437
  Post-visit Follow-up (48 hours post Baseline) | 25.22 (5.11) | 23.04 (6.44)
Statistical Analysis 1: Comparison: Intervention vs Control; Null hypothesis: No difference between study arms in change in mean self-efficacy from Baseline to Post-visit Follow-up; Test type: Superiority; p = 0.011, Mixed Models Analysis — Arm by Time interaction; a priori threshold for statistical significance p<.05; Adjusted for age, purpose of visit, and whether sexually active prior 3 months; random intercepts and slopes over time; clustering by recruitment site; Slope = 1.16, 95% CI 2-sided [0.26 to 2.07] — Arm comparison is Arm 1 (Intervention) minus Arm2 (Control); Time comparison is Post-visit Follow-up minus Baseline
Statistical Analysis 2: Comparison: Intervention; Null hypothesis: No Time difference (Post-visit Follow-up vs. Baseline) in outcome; Test type: Superiority; p < 0.001, Mixed Models Analysis — Post hoc comparison pursuant to significant Arm by Time interaction; a priori threshold for statistical significance p<.05; [statistical method as in outcome 1, analysis 1]; Slope = 1.64, 95% CI 2-sided [1.01 to 2.07] — Time comparison is Post-visit Follow-up minus Baseline
Statistical Analysis 3: Comparison: Control; Null hypothesis: No Time difference (Post-visit Follow-up vs. Baseline) in outcome; Test type: Superiority; p = 0.108, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Slope = 0.48, 95% CI 2-sided [-0.10 to 1.05] — Time comparison is Post-visit Follow-up minus Baseline

2. Primary Outcome: Contraception Use Self-efficacy Scale Score (Aim 1c)
Description: The 3-item attitude scale assessing perceived ability to choose and use contraception was self-administered in an online survey; each item scored on a 0=not at all confident to 10=completely confident scale ; scale score is the sum of the 3 items scores (range 0-30); higher score=greater self-efficacy
Time Frame: Baseline, 3 months, 6 months
Population: All participants for whom a self-efficacy score was recorded at Baseline or at 3 months or at 6 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 690 | 640
Score on a scale
  Pre-Visit Baseline | 23.2 (6.34) | 22.45 (6.72)
  3-month Follow up: number analyzed (Participants) | 282 | 379
  3-month Follow up | 25.22 (4.87) | 23.37 (6.11)
  6-month Follow up: number analyzed (Participants) | 292 | 379
  6-month Follow up | 26.24 (4.38) | 23.44 (5.98)
Statistical Analysis 1: Comparison: Intervention vs Control; Null hypothesis: No difference between study arms in change in mean self-efficacy from Baseline to 3 months or from Baseline to 6 months; Test type: Superiority; p = 0.04, Mixed Models Analysis — Arm by Time interaction; a priori threshold for statistical significance p<.05; [statistical method as in outcome 1, analysis 1]; F statistic:Time X Arm Interaction = 3.23 — df=2,1611; Arm comparison is Intervention - Control; Time comparisons are 3 months - Baseline and 6 months - Baseline and 6 months - 3 months
Statistical Analysis 2: Comparison: Intervention vs Control; Null hypothesis: No difference between study arms in change in mean self-efficacy from Baseline to 3 months; Test type: Superiority; p = .218, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Slope = 0.82, 95% CI 2-sided [-0.48 to 2.11]; Arm comparison is Intervention - Control; Time comparison is 3 months - Baseline
Statistical Analysis 3: Comparison: Intervention vs Control; Null hypothesis: No difference between study arms in change in mean self-efficacy from Baseline to 6 months; Test type: Superiority; p = 0.008, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Slope = 1.58, 95% CI 2-sided [0.38 to 2.77] — Arm comparison is Intervention - Control; Time comparison is 6 months - Baseline

3. Primary Outcome: Percentage of Participants Who Report Using a Non-barrier Method of Birth Control in the Prior 3 Months (Aim 3b)
Description: Recorded via self-administered online survey
Time Frame: Baseline, 3 months, 6 months
Population: All participants who reported what they used to prevent pregnancy in the prior 3 months at Baseline or at 3 months or at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 687 | 650
Participants
  Pre-visit Baseline | 197 | 197
  3-month Follow up: number analyzed (Participants) | 257 | 359
  3-month Follow up | 162 | 161
  6-month Follow up: number analyzed (Participants) | 295 | 379
  6-month Follow up | 185 | 166
Statistical Analysis 1: Comparison: Intervention vs Control; Null hypothesis: No difference between arms in change in percentage of participants using non-barrier method from Baseline to 3 months or to 6 months; Test type: Superiority; p = 0.025, Mixed Models Analysis — Arm by Time Interaction; a priori threshold for statistical significance p<.05; [statistical method as in outcome 1, analysis 1]; F statistic:Time X Arm Interaction = 3.72 — df=2, 1007; Arm comparison is Intervention/Control; Time comparisons are 3 months/Baseline and 6 months/Baseline and 6 months/3 months
Statistical Analysis 2: Comparison: Intervention vs Control; Null hypothesis: No difference between arms in change in percentage of participants using non-barrier method from Baseline to 3 months; Test type: Superiority; p = 0.042, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.29, 95% CI 2-sided [1.04 to 10.36] — Arm comparison is Intervention / Control; Time comparison is 3 months / Baseline
Statistical Analysis 3: Comparison: Intervention vs Control; Null hypothesis: No difference between arms in change in percentage of participants using non-barrier method from Baseline to 6 months; Test type: Superiority; p = 0.005, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.54, 95% CI 2-sided [1.7 to 18.06] — Arm comparison is Intervention / Control; Time comparison is 6 months / Baseline

4. Secondary Outcome: Number of Correct Answers to 7-item Contraception Knowledge Measure (Aim 1a)
Description: The same measure was self-administered in an online survey immediately prior to using the Health-E You app (the intervention) and then immediately after app use. The Health-E You Knowledge Scale is a 7-item true/false format with a range of 0-7, a higher score indicates a better outcome.
Time Frame: Immediate pre-app (Baseline), Immediate post-app (< 1 hour)
Population: Intervention participants who used app
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Intervention: used Healthy-E You app in waiting room prior to clinical visit.
- Control Group Participants: usual care (app not offered)
Arm/Group | Intervention | Control Group Participants
Number analyzed (Participants) | 693 | 0
Scores on a scale
  Pre-App Knowledge Scale | 3.31 (1.61) |
  Post-App Knowledge Scale: number analyzed (Participants) | 549 | 0
  Post-App Knowledge Scale | 4.94 (1.74) |
Statistical Analysis 1: Comparison: Intervention; Null hypothesis: No change in contraception knowledge from immediate pre-app to immediate post-app among Intervention group participants; Test type: Superiority; p < 0.001, Mixed Models Analysis — Time main effect; a priori threshold for statistical significance p <.05; [statistical method as in outcome 1, analysis 1]; Slope = 1.62, 95% CI 2-sided [1.43 to 1.82] — Time comparison is post-app minus pre-app

5. Secondary Outcome: Percentage of Participants Who Report Discussing Birth Control With Health Care Provider at Visit (Aim 2b)
Description: The single yes/no item was self-administered in an online survey
Time Frame: Post-visit Follow-up (48 hours after Baseline)
Population: All participants who completed the item at Post-visit Follow-up (48 hours post-visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 320 | 436
Participants | 285 | 301
Statistical Analysis 1: Comparison: Intervention vs Control; Null hypothesis: No difference between study arms in percentage of participants who discussed birth control with health care provider at visit; Test type: Superiority; p = 0.055, Regression, Logistic — Arm main effect; a priori threshold for statistical significance p<.05; Adjusted for age, purpose of visit, and whether sexually active prior 3 months; clustering by recruitment site; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.98 to 5.01] — Arm comparison is Arm 1 (Intervention) / Arm2 (Control)

6. Secondary Outcome: Percentage of Participants Who Receive or Make an Appointment to Receive or Receive a Prescription for a Non-barrier Method (Aim 3a)
Description: Recorded via self-administered online survey
Time Frame: Post-visit Follow-up
Population: All participants who answered the appropriate items at Post-visit Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 319 | 436
Participants | 236 | 221
Statistical Analysis 1: Comparison: Intervention vs Control; Null hypothesis: No difference between study arms in percentage of participants who receive/make appointment/get prescription for a non-barrier method; Test type: Superiority; p = 0.227, Regression, Logistic — Arm main effect; a priori threshold for statistical significance p<.05; Adjusted for age, purpose of visit, and whether sexually active prior 3 months; clustering by recruitment site; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.73 to 3.78] — Arm comparison is Arm 1 (Intervention) / Arm2 (Control)

7. Secondary Outcome: Post-study Assessment of Providers' Rating of How the Health-E You APP Improves the Effectiveness of the Clinical Encounter for Patients: App Helps Patients Engage in Contraception Decision Making (Aim 2a1)
Description: Provider ratings of whether the App improves the effectiveness of the clinical encounter for patients, using a Likert scale (options 1- strongly disagree to 5- strongly agree); then dichotomized into agrees versus neutral/disagrees.
Time Frame: Post-study completion
Population: Providers seeing patients for care in Health-E You Intervention Clinics
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Providers: Clinical providers in Health-E You Intervention Clinics
Arm/Group | Clinical Providers
Number analyzed (Participants) | 12
Participants
  Agree helps patients in decision making | 10
  Neutral/disagree helps in decision making | 2

8. Secondary Outcome: Post-study Assessment of Provider Ratings of Whether the Health-E You APP Helps Clinicians Provide Individually Tailored Discussion of Contraception Options (Aim 2a2)
Description: Provider ratings of whether the App helps clinicians provide more individually tailored discussion of contraception options, using a Likert scale (options 1- strongly disagree to 5- strongly agree); then dichotomized into agrees versus neutral/disagrees.
Time Frame: Post-study completion
Population: Clinical providers in Health-E You Intervention Clinics
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Providers
Number analyzed (Participants) | 12
Participants
  Agrees it helps clinicians | 9
  Neutral/disagrees it helps clinicians | 3

9. Secondary Outcome: Post-study Assessment of Provider Ratings of Whether the Health-E You APP Improves the Effectiveness of the Clinical Encounter by Integrating Reproductive Health Into All Visits (Aim 2a3)
Description: Provider ratings of whether the App improves effectiveness of the clinical encounter by integrating reproductive health into all visits, using a Likert scale (options 1- strongly disagree to 5- strongly agree); then dichotomized into agrees versus neutral/disagrees.
Time Frame: Post-study completion
Population: Clinical providers in Health-E You Intervention Clinics
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Providers
Number analyzed (Participants) | 12
Participants
  Agree it helps integrate reproductive care | 6
  Neutral/disagrees it helps | 6

10. Secondary Outcome: Post-study Assessment of Provider Ratings of Whether the Health-E You APP Makes Clinic Schedule Run Behind (Aim 2a4)
Description: Provider ratings of whether the App makes clinic schedules run behind, using a Likert scale (options 1- strongly disagree to 5- strongly agree); then dichotomized into agrees versus neutral/disagrees.
Time Frame: Post-study completion
Population: Clinical providers in Health-E You Intervention Clinics
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Providers
Number analyzed (Participants) | 12
Participants
  Agrees App makes clinic schedules run behind | 0
  Neutral/disagree APP makes schedules run behind | 12

11. Secondary Outcome: Adolescent Assessment of Health-E You App Benefits: Helped me Choose a Birth Control Method (Aim 2a5)
Description: Response to query about agreement with App benefits on 5 point Likert scale (1-strongly disagree to 5- strongly agree); dichotomized into agree versus neutral/disagree
Time Frame: Immediate Follow-up
Population: Intervention group adolescents
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Intervention Arm- completed Health-E You App
Arm/Group | Intervention
Number analyzed (Participants) | 287
Participants
  Agree APP helped choose method | 198
  Neutral/disagree APP helped choose method | 89

12. Secondary Outcome: Adolescent Assessment of Health-E You App Benefits: Gave me Useful Information About Birth Control (Aim 2a6)
Description: as for outcome 11
Time Frame: Immediate Follow-up
Population: Intervention group adolescents
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 287
Participants
  Agree APP gave useful birth control information | 250
  Neutral/disagree APP gave useful information | 37

13. Secondary Outcome: Adolescent Assessment of Health-E You App Benefits: Helped me Talk With my Health Care Provider About Birth Control (Aim 2a7)
Description: as for outcome 11
Time Frame: Immediate Follow-up
Population: Intervention group adolescents
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 287
Participants
  Agree it helped me talk with provider | 192
  Neutral/disagree it helped me talk with provider | 95

14. Secondary Outcome: Adolescent Assessment of Health-E You App Benefits: Improved the Quality of my Visit With my Health Care Provider (Aim 2a8)
Description: as for outcome 11
Time Frame: Immediate Follow-up
Population: Intervention group adolescents
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 287
Participants
  Agree it helped quality of visit with provider | 200
  Neutral/disagree it helped quality of visit | 87

ADVERSE EVENTS:
Time Frame: This study was of minimal risk to participants. Participants were enrolled in the study for a total of 6 months from completion of baseline to end of follow-up. Adverse event data was collected during this time frame.
Description: There were no adverse events that occurred during this study. This study was of minimal risk to participants.
Arm/Group | Health-E You Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/693 | 0/667
Serious Adverse Events (participants affected / at risk) | 0/693 | 0/667
Other Adverse Events (participants affected / at risk) | 0/693 | 0/667

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT02847858/Prot_SAP_000.pdf